CLINICAL TRIAL: NCT06904820
Title: Acceptability and Feasibility of Simultaneous Screening for Viral Hepatitis B, C and HIV Among Drug Users and Vulnerable Populations, in Non-conventional Structures "Outside the Walls" by Dual Screening Method RTDs and FibroScan®
Acronym: SCANVIRE2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI24_0061 (SCANVIRE2)
Record Dates: First submitted 2025-02-21; First posted 2025-04-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: Viral Hepatitis
Keywords: HCV; eradication; marginalized patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The "Scanvir" concept aims to achieve barriers to HCV screening and treating of marginalized patients. The concept is applicable to other various populations and territories and should effectively improve HCV patient's health outcomes. The main objective of the SCANVIR project was to evaluate the feasibility, acceptability and reproducibility of a "test, treat and cure" strategy for PWIDs and vulnerable populations during dedicated days in addiction care centers.

DETAILED DESCRIPTION:
According to the French recommendations, eliminating hepatitis C virus by 2025 could be a realistic public health goal in this country. A total of 71,466 patients had treatment initiation between 2015 and 2019. It is estimated that 100 000 people are still infected in 2019.

To meet these ambitious objectives, effective screening policies should be intensified and access to treatment promoted through new care strategies for patients who escape the usual care pathways i.e. people who inject drugs (PWIDs), prisoners, migrants and vulnerable populations.

PWIDs represent a large proportion of patients to be screened and treated. It's still not possible to accurately evaluate the number of drug users who are infected with HCV (45 000 people estimated).

Drug users sharing needles and syringes have poor access to treatment. Dealing with PWIDs in addiction care centers (CSAPA and CAARUD in France) is one way to promote HCV testing, and to keep them in the care pathway. This population requires dedicated models that reduce barriers to care: harm reductions policies, access to therapy in real time and follow-up for the detection of reinfection. So the investigator designed and applied a new innovative concept to test, treat and cure PWIDs in their own environment, called the SCANVIR program, initially tested in four French departments with a regional and now national extension.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 and over
* Patient frequenting an unconventional structure "outside the walls" or referred by a professional in the care sector
* Patient not opposed to research

Exclusion Criteria:

* Age under 18
* Patient opposed to research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: drug users and vulnerable populations in non-conventional structures
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2035-06-05 (Estimated); Study Completion 2035-06-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the acceptability and the feasibility of simultaneous screening for viral hepatitis B, C and HIV among drug users and vulnerable populations in non-conventional structures using a triple method with RTD and FibroScan® and GeneXpert®. | from enrollment to the end of the subject participation at the end of the day
  Feasibility will be assessed by the number of days and the number of participants in all sessions.
  the acceptability of TROD and/or Fibroscan will be assessed by the number and proportion of double screenings (TROD and/or Fibroscan) performed in relation to the number of screenings offered

SECONDARY OUTCOMES:
Reinforce screening for hepatitis B (HBV), hepatitis Delta (HDV) and HIV, | from enrollment to the end of the subject participation at the end of the day
  Number and proportion of patients who accepted immediate consultation with the hepatologist,
Reinforce education to prevent the risk of viral transmission, | from enrollment to the end of the subject participation at the end of the day
  Number and proportion of patients who accepted risk prevention education by the nurse
Encourage HBV vaccination, | from enrollment to the end of the subject participation at the end of the day
  Number of HBV vaccinations offered,
Evaluate the feasibility of PCR (GeneXpert/Buvard), | from enrollment to the end of the subject participation at the end of the day
  Number of GeneXpert PCRs performed, Number of PCRs performed on blotting paper,
Reinforce education to prevent the risk of viral transmission, | from enrollment to the end of the subject participation at the end of the day
  Number and proportion of patients who have accepted risk prevention education from the nurse,
Provide social support, | from enrollment to the end of the subject participation at the end of the day
  Number of patients who received social support,
Offer rapid treatment to HCV-positive patients in precarious situations, | from enrollment to the end of the subject participation at the end of the day
  Absolute number and proportion of patients treated or not maintained in care,
Assess associated co-morbidities: alcohol, cannabis, drug misuse, associated psychiatric pathologies, | from enrollment to the end of the subject participation at the end of the day
  Number of patients with one or more risk factors for chronic liver disease, whether or not associated with chronic viral hepatitis or HIV infection: alcohol, metabolic syndrome, cannabis, drugs detected by FibroScan ®.

CONTACTS AND LOCATIONS:
Overall Officials: marilyne DEBETTE-GRATIEN, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges University Hospital, Limoges, France